CLINICAL TRIAL: NCT06475092
Title: Relation Between Muscle Mass, Total Body Fat, Visceral Fat, Waist Hip Ratio and Sleeping Hours in Patient With Nonspecific Back Pain
Status: Completed | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Ababa, lecturer of internal physical therapy, Ahram Canadian University
Other Study IDs: P.T-ORT 06/2024-546
Record Dates: First submitted 2024-06-11; First posted 2024-06-26 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Back Pain; Sleep
MeSH Terms: conditions — Obesity; Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Tanita device — bioelectric impedance analysis
  Other Names: tap measurement

SUMMARY:
Objective: To find out if there are a relation between muscle mass, total body fat, visceral fat, waist hip ratio and sleeping hours in patient with nonspecific back pain.

Design: Cross sectional study. Subjects: 30 male and female patients with age ranged from 25 to 40 years old diagnosed as nonspecific low back pain will participate in this study.

Main measures: the Outcome measures will be including the assessment of muscle mass, total body fat, visceral fat, waist hip ratio and sleeping hours.

Results: The results will be analyzed via co relation test.

DETAILED DESCRIPTION:
Objective: To find out if there are a relation between muscle mass, total body fat, visceral fat, waist hip ratio and sleeping hours in patient with nonspecific back pain.

methods:

* tatinia bioelectric impedance device used for measurement of muscle mass total body fat and visceral fat
* waist hip ratio measured by tape measurement The waist-hip ratio or waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement (W⁄H).

participants 30 male and female patient will participate in this study

ELIGIBILITY:
Inclusion Criteria:

* •adulthood with low back pain

  * Their ages will range from 20-40 years old.
  * All of them suffer from mild to moderate degree of low back pain.
  * The subjects complain from low back pain for 1 month ago

Exclusion criteria:

Exclusion criteria were a history of any of the following condition:

* inflammatory diseases or any rheumatic disorders,
* a history of vertebral fractures
* surgical spinal fixation.
* •any neurological disorders like MS

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 male and female patient, Their ages will range from 20-40 years old. All of them suffer from mild to moderate degree of low back pain. and they complain from low back pain for 1 month ago
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Tanita device will be used for measurement of total body fat , muscle mass and visceral fat | baseline
  bioelectric impedance analysis device will be used for assessment of total body fat ,muscle mass and viseral fat
Waist hip ratio will be measured by tape measurement | base line
  The waist-hip ratio or waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement (W⁄H).

CONTACTS AND LOCATIONS:
Locations (1):
- Ahram Canadian university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No